CLINICAL TRIAL: NCT03750604
Title: Central Obesity With Relation in OAB: Is it a Matter of Size or Fat Activity?. Prospective Controlled Trial
Brief Title: Central Obesity in Cases of OAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohamed Abdelbaset, principal investigator, Mansoura University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: obesity in OAB
Record Dates: First submitted 2018-11-09; First posted 2018-11-23 (Actual); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: Urologic Diseases; Overactive Bladder Syndrome; Obesity, Abdominal
Keywords: abdominal obesity; OAB
MeSH Terms: conditions — Urologic Diseases; Obesity, Abdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients with OAB (Active Comparator): Patients were asked to fill (OABSS) for more accurate evaluation of bothersome degree. Waist Circumference is evaluated. The surface area of subcutaneous fat (S) and visceral (V) is calculated using slices between L4-L5 and umbilicus according to CT detection fat methods Also bladder wall thickness was calculated by measuring average bladder wall thickness at three different levels. Subcutaneous fat to visceral fat ratio was calculated. Assays for serum total and high-density lipoprotein cholesterol (HDL-C) and triglyceride (TG) levels were performed in the hospital's chemistry laboratory with an autoanalyzer. VAI was calculated for females as this formula like the previous study.
  VAI: WC/ [36.58 + (1.89 × BMI)] × TG/0.81 × 1.52/HDL.
  And in males:
  VAI: WC / [39.68 + (1.88 x BMI)] x TG/ 1.03 x 1.31/ HDL
  Interventions: Diagnostic Test: visceral fat obesity (surface area and function)
- normal variants healthy without symptoms (Placebo Comparator): WC is evaluated crest. The surface area of subcutaneous fat (S) and visceral (V) is calculated using slices between L4-L5 and umbilicus according to ct detection fat methods Also bladder wall thickness was calculated by measuring average bladder wall thickness at three different levels. Subcutaneous fat to visceral fat ratio was calculated. Assays for serum total and high-density lipoprotein cholesterol (HDL-C) and triglyceride (TG) levels were performed in the hospital's chemistry laboratory with an autoanalyzer. VAI was calculated for females as this formula like the previous study.
  VAI: WC/ [36.58 + (1.89 × BMI)] × TG/0.81 × 1.52/HDL. And in males:VAI: WC / [39.68 + (1.88 x BMI)] x TG/ 1.03 x 1.31/ HDL
  Interventions: Diagnostic Test: visceral fat obesity (surface area and function)

INTERVENTIONS:
Diagnostic Test: visceral fat obesity (surface area and function) — WC is evaluated at the midpoint between the lower border of the rib cage and the iliac crest. The surface area of subcutaneous fat (S) and visceral (V) is calculated using slices between L4-L5 and umbilicus according to ct detection fat methods Also bladder wall thickness was calculated by measuring average bladder wall thickness at three different levels.
  Subcutaneous fat to visceral fat ratio was calculated. Assays for serum total and high-density lipoprotein cholesterol (HDL-C) and triglyceride (TG) levels were performed in the hospital's chemistry laboratory with an autoanalyzer. VAI was calculated for females as this formula like the previous study.
  VAI: WC/ [36.58 + (1.89 × BMI)] × TG/0.81 × 1.52/HDL.
  And in males:
  VAI: WC / [39.68 + (1.88 x BMI)] x TG/ 1.03 x 1.31/ HDL WC: waist circumference, BMI: body mass index, TG: triglyceride, HDL: high-density lipoprotein

SUMMARY:
Obesity is not a homogeneous condition and that the regional distribution of adipose tissue is important to understanding the relation of obesity to disturbances in glucose and lipid metabolism. Central abdominal fat is composed of abdominal subcutaneous fat and visceral fat. Regional distribution appears to be an important indicator for metabolic alterations since an inconstant correlation between body mass index (BMI) and these disturbances have been found. Visceral obesity is associated with increased adipocytokine production, proinflammatory activity, deterioration of insulin sensitivity, increased risk of developing diabetes, "high-triglyceride/low-HDL cholesterol dyslipidemia," hypertension and atherosclerosis. It might be more precise to divide central abdominal fat into subcutaneous(S) and visceral (V) fat surface area and volume and even ratio (S/V); risk factors for cardiovascular disease, particularly those related to glucose and lipid metabolism and hypertension, being>0.4; with evaluation of visceral fat functionality by visceral adiposity index (VAI) with integration with lipid profile. Adding bladder wall thickness with perivesical fat as a factor may impair bladder function and contribute to dysregulation. The data on the association between central adiposity with OAB symptoms and Urodynamics is not mature.

DETAILED DESCRIPTION:
Overactive bladder (OAB) is defined by international continence society (ICS) as urinary urgency with or without incontinence often associated with frequency and nocturia. As a chronic, unbearable condition, OAB has a deeply negative impact on QoL, including social, physical, psychological, occupational and sexual domains. Overactive bladder (OAB) is a highly prevalent symptom complex that is estimated to affect 12.8% of women and 10.8% of men.

The underlying pathophysiological mechanism of OAB and DO is poorly understood. It is thought that not only the detrusor muscle but also urothelium, peripheral afferent terminals, and pelvic blood vessels may play a role.

More recently, overweight and central obesity was found to be an independent risk factor for overactive bladder (OAB) in women. The most likely explanation is the occurrence of chronic inflammation in the bladder indicated by increased urinary chemokines. Adipocytes surrounding the human bladder can be affected, thus leading to inflammation and triggering OAB symptoms. Other authors showed that OAB is associated with increased BMI and increase of waist circumference at the upper end of the adiposity distribution for both men and women.

Obesity is not a homogeneous condition and that the regional distribution of adipose tissue is important to understanding the relation of obesity to disturbances in glucose and lipid metabolism. Central abdominal fat is composed of abdominal subcutaneous fat and visceral fat. Regional distribution appears to be an important indicator for metabolic alterations since an inconstant correlation between body mass index (BMI) and these disturbances have been found. Visceral obesity is associated with increased adipocytokine production, proinflammatory activity, deterioration of insulin sensitivity, increased risk of developing diabetes, "high-triglyceride/low-HDL cholesterol dyslipidemia," hypertension and atherosclerosis.

Away from that anthropometric measures as BMI, waist circumference (WC), waist to hip ratio (WHR) are crude measures for adiposity. WHR has been advocated as a measure of central obesity because BMI does not describe the distribution of obesity. This measurement, however, was found to be associated with SUI but not with OAB or mixed urinary incontinence, further suggesting a non-mechanical mechanism for OAB in obese women. WC is a major clinical parameter used for the indirect evaluation of increased visceral fat, In addition, WC showed shared variance with visceral adipose fat up to 75% (42) (38). Nevertheless, WC alone does not help in distinguishing between subcutaneous and visceral fat mass.

So, it might be more precise to divide central abdominal fat into subcutaneous(S) and visceral (V) fat surface area and volume and even ratio (S/V); risk factors for cardiovascular disease, particularly those related to glucose and lipid metabolism and hypertension, being>0.4; with evaluation of visceral fat functionality by visceral adiposity index (VAI) with integration with lipid profile. Adding bladder wall thickness with perivesical fat as a factor may impair bladder function and contribute to dysregulation.

The data on the association between central adiposity with OAB symptoms and Urodynamics is not mature. So, the investigators intend to conduct this study evaluating the surface area of both subcutaneous and visceral fat and its functionality with incorporation with lipid profile and bladder wall thickness and perivesical fat.

ELIGIBILITY:
Inclusion Criteria:

* patients with OAB between 18 and 40 years old.
* normal variant healthy donor as a control.

Exclusion Criteria:

* Patients who have any of the following:

  * Age less than 18 or more than 40 years old
  * Neurogenic detrusor overactivity
  * evidence of obstructed flow in absence of prolapse
  * mixed urinary incontinence
  * associated urethral pathology, e.g. Urethral diverticulum
  * Associated bladder pathology e.g. fistula, active urinary tract infection as evidenced by positive urine culture
  * previous exposure for anticholinergics or BTX-A injection.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 250 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
relation between visceral fat and and severity of OAB symptoms. | 2 years
  using OAB symptoms scores(OABSS) with total score 15(mild<5,mod (5-10),sever>10) in relation to visceral fat surface area in cm2 by NCCT measurement.
Relation of OAB symptoms to visceral fat function | 2 years
  using of OABSS total score 15(mild<5, mod(5-10), sever>10) to visceral fat function (VAI)(VAI: WC/ [36.58 + (1.89 × BMI)] × TG/0.81 × 1.52/HDL. And in males:VAI: WC / [39.68 + (1.88 x BMI)] x TG/ 1.03 x 1.31/ HDL)